CLINICAL TRIAL: NCT00825344
Title: A Randomized Controlled Study Evaluating Pre-operative Etanercept on the Severity of Postoperative Pain After Inguinal Hernia Surgery.
Brief Title: Preoperative Etanercept Before Inguinal Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); John P. Murtha Neuroscience and Pain Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WU08-6987
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Inguinal Hernia; Postoperative Pain
Keywords: postoperative pain; inguinal hernia; chronic postsurgical pain; cytokine; preemptive analgesia; patients with inguinal hernia scheduled for surgery
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Etanercept; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Etanercept 50 mg preoperatively
  Interventions: Drug: Etanercept
- 2 (Placebo Comparator): Subcutaneous saline preoperatively
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Etanercept — 50 mg subcutaenous preoperatively
  Arms: 1
Drug: Saline — Given subcutaneously preoperatively
  Arms: 2

SUMMARY:
Inguinal hernia repair is one of the most frequently performed operations in young men. Persistent pain after inguinal surgery represents a significant cause of disability, occurring in between 15%-35% of cases. In a majority of these patients, their groin pain persisted after a previous hernia repair. The main type of chronic postsurgical pain is neuropathic, caused by injured nerves. One of the principal components in the pathophysiology of postsurgical pain is cytokines, specifically tumor necrosis factor (TNF). In animal studies, injecting TNF inhibitors before nerve injury can reduce pain behaviors and neuropathology. Finding a way to reduce the incidence of postsurgical pain after hernia repair could enhance function, and reduce the need for opioids and other analgesics. The investigators intend to conduct the first randomized, controlled study evaluating whether preemptive administration of a tumor necrosis inhibitor can reduce postoperative pain and opioid consumption after hernia repair. This is important because the degree and intensity of postsurgical pain is a major predictor for the development of chronic postsurgical pain.

DETAILED DESCRIPTION:
76 patients with an inguinal hernia scheduled for surgical repair will be randomized in a 1:1 ratio to receive either subcutaneous etanercept or saline before skin incision. The study will be double-blind (i.e. neither the surgeon, anesthesiologist, nor the person administering the injection will know which group they were assigned to). Group I will receive 50 mg of subcutaneous etanercept mixed in 1 ml sterile water 90-120" before skin incision. Group II will receive 1 ml of sterile water 90-120" before skin incision. The anesthesia and surgical procedures will be standardized. For the next 24 hours, patients will keep a q4 hour pain diary recording their average pain on a 0-10 numerical rating scale. They will also record the number of Percocet tablets they took. All patients will be seen 1 month after their surgery, where their average pain score, work status, and analgesic intake (if any) will be recorded. Patients will then be followed with a telephone follow-up 3, 6 and 12-months post-procedure, where the same variables will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrable hernia evident using ultrasound, computed tomography, or on physical exam.
2. Pt scheduled for unilateral inguinal hernia repair.
3. Symptoms present for < 6 months.

Exclusion Criteria:

1. Non-elective surgery.
2. Previous hernia repair at the same site, or surgery near the site of the hernia.
3. Demyelinating neurological disease.
4. Current or recent (< 6 years) history of substance abuse.
5. Pregnancy, which will be ruled out by a urine pregnancy test in women of childbearing age.
6. Pre-existing untreated psychiatric condition that could preclude an optimal treatment response (e.g. untreated posttraumatic stress disorder).
7. Unstable medical condition (e.g. unstable angina or congestive heart failure or severe).
8. Rheumatoid arthritis, or other systemic conditions that might respond to TNF inhibitors.
9. Pt is immunosuppressed or is taking other drugs (e.g. corticosteroids) that might suppress the immune system.
10. Systemic infection.
11. Any opioid analgesics within 48 hours of skin incision.
12. Any use of tricyclic antidepressants, serotoninin-norepinephrine reuptake inhibitors, or anticonvulsants within 72 hours of skin incision.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rehrig, MD, Study Chair — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Cheek CM, Black NA, Devlin HB, Kingsnorth AN, Taylor RS, Watkin DF. Groin hernia surgery: a systematic review. Ann R Coll Surg Engl. 1998;80 Suppl 1:S1-80. PMID 11432408
- [Background] Franneby U, Sandblom G, Nordin P, Nyren O, Gunnarsson U. Risk factors for long-term pain after hernia surgery. Ann Surg. 2006 Aug;244(2):212-9. doi: 10.1097/01.sla.0000218081.53940.01. PMID 16858183
- [Background] Ferzli GS, Edwards E, Al-Khoury G, Hardin R. Postherniorrhaphy groin pain and how to avoid it. Surg Clin North Am. 2008 Feb;88(1):203-16, x-xi. doi: 10.1016/j.suc.2007.10.006. PMID 18267170
- [Background] Sommer C, Kress M. Recent findings on how proinflammatory cytokines cause pain: peripheral mechanisms in inflammatory and neuropathic hyperalgesia. Neurosci Lett. 2004 May 6;361(1-3):184-7. doi: 10.1016/j.neulet.2003.12.007. PMID 15135924

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept 50 mg preoperatively
  Etanercept : 50 mg subcutaenous preoperatively
- Saline: Subcutaneous saline preoperatively
  Saline : Given subcutaneously preoperatively
Period: Overall Study
Arm/Group | Etanercept | Saline
Started | 34 | 43
Completed | 33 | 42
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Etanercept 50 mg preoperatively
  Etanercept : 50 mg subcutaenous preoperatively
- Group 2: Subcutaneous saline preoperatively
  Saline : Given subcutaneously preoperatively
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 34 | 43 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 8 | 18 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (3.1) | 58.4 (2.8) | 57.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 31 | 40 | 71
Region of Enrollment [Number; unit: participants]
  United States | 34 | 43 | 77

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale Pain Score
Description: 0-10 pain score through 24-hours post-surgery. 0 is no pain and 10 is the worse pain imaginable. The primary outcome reported measure is the average of 4 scores, each comprised of 6-hour time intervals during the 24hour period.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Saline
Number analyzed (Participants) | 34 | 43
units on a scale | 3.3 (1.9) | 3.9 (2.3)

2. Secondary Outcome: Analgesic Usage
Description: Number of oxycodone/ acetaminophen tablets consumed through 24 hours post-surgery
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Etanercept | Saline
Number analyzed (Participants) | 34 | 43
tablets | 4.0 (2.8) | 5.8 (4.2)

3. Secondary Outcome: Chronic Post-surgical Pain
Description: Patients with persistent post-surgical pain
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Etanercept | Saline
Number analyzed (Participants) | 33 | 42
participants | 5 | 5

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/43
Other Adverse Events (participants affected / at risk) | 0/34 | 0/43

LIMITATIONS AND CAVEATS:
Only one type of surgery studied; more males than females enrolled (function of military treatment facility and type of population)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No